CLINICAL TRIAL: NCT01192529
Title: Clinical Evaluation of an Specific Diet for People With Dementia Disease
Brief Title: Evaluation of a Diet in Patients With Senile Dementia
Acronym: SUPRESSI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vegenat, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: VEGENAT-SUPR; SUPRESSI2010-PROYECTO CDTI (Other: VEGENAT, S.A.)
Record Dates: First submitted 2010-08-30; First posted 2010-09-01 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2011-02

CONDITIONS: Alzheimer's Disease; Parkinson's Disease; Senile Dementia
Keywords: Senile; Dementia; Neurodegenerative; Supressi; Specific diet; Cognitive Status; Memory; Malnutrition; Parkinson; Alzheimer
MeSH Terms: conditions — Alzheimer Disease; Parkinson Disease; Dementia; Malnutrition

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Group (Experimental): In addition to their daily diet, patients of this group will receive 400 ml per day of "Supressi" nutritional supplement
  Interventions: Dietary Supplement: Supressi. T-Diet plus Range
- Control Group (Active Comparator): In addition to their daily diet, patients of this group will receive 400 ml per day of "T-Diet plus High Protein" product
  Interventions: Dietary Supplement: High Protein. T-Diet plus Range

INTERVENTIONS:
Dietary Supplement: Supressi. T-Diet plus Range — Supressi is a complete high protein and moderated high energy oral nutrition supplement, indicated for the dietary management of patients with neurodegenerative diseases and related malnutrition.
  Experimental group patients will receive, 2 packs per day (Tetra brik aseptic)of 200 ml for 6 months.
  Other Names: VEG001
  Arms: Experimental Group
Dietary Supplement: High Protein. T-Diet plus Range — T-Diet plus High Protein is a complete high protein and moderated high energy oral nutrition supplement, indicated for the dietary management of patient with related malnutrition and with increased protein requirements.
  Other Names: VEG002
  Arms: Control Group

SUMMARY:
The most common symptoms associated to senile dementia disease are confusion about schedules, hyperactivity... In this sense, these patients have frequently poor nutrition, resulting in malnutrition problems or malnutrition high risk.

DETAILED DESCRIPTION:
The purpose of this study is to assess if the daily intake of a specific nutritional supplement versus a non specific supplement one is related to malnutrition or malnutrition risk reduction and contributes to an improvement in cognitive and functional parameters in patients with senile dementia.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 70 years with neurologist or geriatrician dementia diagnosis (Alzheimer's disease, Parkinson's or mixed), with mild or moderate cognitive impairment degree (Between 24 and 14 MMSE).
* Patients with or at malnutrition risk (Mini Nutritional Assessment screening positive)

Exclusion Criteria:

* Patients with decompensated kidney failure, creatine and/or bilirubin greater than 2, uric acid higher than 8 mg/dl, and glomerular filtration under 60 ml/minute.
* Patients with Diabetes mellitus poorly controlled (Glycemia > 200 mg/dl)
* Patients with decompensated hypertension.
* Patients with pharmacological treatment or consuming supplements containing specific supplementation of experimental product (omega 3 and/or vitamins supplements).
* Post-stroke vascular dementias.
* Do not achieve any inclusion criteria.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2010-10; Primary Completion 2012-09 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Nutritional and cognitive status in elderly people | 1 year
  The evaluation include: Nutritional evaluation, Improvement of Anthropometric and Biochemical parameters evaluation in relation to patient malnutrition, Patient's cognitive status evaluation (Folstein's MMSE and GDS scale), Functional and psychopathological aspects evaluation (blessed Scale), Global Impresion of Change Evaluation(CIBIC plus Scale), Quality of life evaluation (Short Form 36 questionaire), Memory Evaluation (Rey Auditory Learning Test), Appearance of gastrointestinal events evaluation, Diet and Intake acceptance evaluation.

SECONDARY OUTCOMES:
Biochemical parameters measure | 8 months
  Fatty acid profile of plasma and erythrocytes, plasma levels of some proinflammatory cytokines and b-amyloid, genotyped, oxidative stress determination, total proteins determination, total lymphocytes, albumin, pre-albumin, transferrine, Reactive C protein (RCP), homocystein, total cholesterol, plasma level of glucose, Homeostasis Model Assessment and Renal function.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio J Pérez de la Cruz, MD PhD, Principal Investigator — Clinical Nutrition and Dietetic Unit, University Hospital Virgen de las Nieves; Ángel Gil Hernández, PhD, Principal Investigator — Department of Biochemistry and Molecular Biology II. University of Granada; Adrián Arés Luque, MD, Principal Investigator — Neurological Unit, Complejo Asistencial de León
Locations (3):
- Spain (3):
  - Clinical Nutrition and Dietetic Unit, University Hospital Virgen de las Nieves, Granada, Granada
  - Department of Biochemistry and Molecular Biology II. University of Granada, Granada, Granada
  - Neurological Unit, Complejo Asistencial de León, León, León